CLINICAL TRIAL: NCT04454658
Title: A Phase 1b Study Of ABBV-744 Alone Or In Combination With Ruxolitinib Or Navitoclax In Subjects With Myelofibrosis
Brief Title: Safety and Tolerability Study of Oral ABBV-744 Tablet Alone or in Combination With Oral Ruxolitinib Tablet or Oral Navitoclax Tablet in Adult Participants With Myelofibrosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-247; 2020-001225-32 (EudraCT Number)
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Myelofibrosis (MF)
Keywords: ABBV-744; Navitoclax; Ruxolitinib; ABT-263; Cancer; Myelofibrosis; MF
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasms | interventions — ABBV-744; navitoclax; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Segment A: ABBV-744 Dose Identification and Optimization (Experimental): Participants who have been previously treated with Janus Kinase inhibitor(s) (JAKi) and stopped such therapy, will receive different dosing regimens and schedules of ABBV-744 to identify the safe dosing regimen and schedule.
  Interventions: Drug: ABBV-744
- Segment A: ABBV-744 Monotherapy (Experimental): Participants will receive the identified safe dosing regimen of ABBV-744 as monotherapy.
  Interventions: Drug: ABBV-744
- Segment B: Ruxolitinib + ABBV-744 "Add on" Therapy (Experimental): Participants whose disease (myelofibrosis) is inadequately controlled by ongoing ruxolitinib therapy will receive ruxolitinib and ABBV-744 as "add-on" therapy.
  Interventions: Drug: ABBV-744; Drug: Ruxolitinib
- Segment C: ABBV-744 + Navitoclax (Experimental): Participants who have previously been exposed to JAKi, and stopped such therapy, will receive ABBV-744 and navitoclax.
  Interventions: Drug: ABBV-744; Drug: Navitoclax
- Segment D: ABBV-744 + Ruxolitinib (Experimental): Participants who have never received JAKi will receive ABBV-744 and ruxolitinib.
  Interventions: Drug: ABBV-744; Drug: Ruxolitinib

INTERVENTIONS:
Drug: ABBV-744 — Tablet; Oral
Drug: Navitoclax — Tablet; Oral
  Other Names: ABT-263
  Arms: Segment C: ABBV-744 + Navitoclax
Drug: Ruxolitinib — Tablet; Oral
  Arms: Segment B: Ruxolitinib + ABBV-744 "Add on" Therapy; Segment D: ABBV-744 + Ruxolitinib

SUMMARY:
Myelofibrosis (MF) is a bone marrow illness that affects blood-forming tissues in the body. MF disturbs the body's normal production of blood cells, causing extensive scarring in the bone marrow. This leads to severe anemia, weakness, fatigue, and an enlarged spleen. The purpose of this study is to see how safe and tolerable ABBV-744 is, when given alone, and in combination with ruxolitinib or navitoclax, for adult participants with MF.

ABBV-744 is an investigational drug being developed for the treatment of MF. The study has 4 segments - A, B, C, and D. In Segment A, the safe dosing regimen of ABBV-744 is identified and then, given alone as monotherapy. In Segment B, C, and D, combination therapies of ABBV-744 with either ruxolitinib or navitoclax are given. Adult participants with a diagnosis of MF will be enrolled. Around 130 participants will be enrolled in 60 sites worldwide.

In Segment A, participants will receive different doses and schedules of oral ABBV-744 tablet to identify safe dosing regimen. Additional participants will be enrolled at the identified monotherapy dosign regimen. In Segment B, participants will receive oral ruxolitinib and ABBV-744 will be given as "add-on" therapy. In Segment C, participants will receive ABBV-744 and oral navitoclax. In Segment D, participants will receive ABBV-744 and ruxolitinib. Participants will receive treatment until disease progression or the participants are not able to tolerate the study drugs.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of treatment will be checked by medical assessments, blood and bone marrow tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory values indicative of adequate bone marrow, renal, and hepatic function meeting protocol criteria.
* Completion of the Myelofibrosis System Assessment Form (MFSAF) on at least 4 out of the 7 days prior to Day 1 with at least 2 symptoms with a score >=3 or a total score of >=10.
* Documented diagnosis of intermediate or high-risk primary myelofibrosis (PMF), post-polycythemia vera MF (PPV-MF) or post-essential thrombocytopenia MF (PET-MF) as defined by the World Health Organization (WHO).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of <= 2.
* Intermediate - 2, or High-Risk disease as defined by the Dynamic International Prognostic Scoring System (For Segment A only, Intermediate - 1 with palpable splenomegaly >=5 centimeters [cm] below costal margin are also eligible).
* Splenomegaly defined as spleen palpation measurement >= 5 cm below costal margin or spleen volume >= 450 cubic cms as assessed by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) scan (for Segments A and C, baseline spleen assessment must be obtained > 7 days after discontinuation of most recent Myelofibrosis (MF) therapy. If possible, this assessment should occur within 10 days of Cycle 1 Day 1).

Segment-Specific Prior Therapy Criteria:

* Segment A:

  * Prior exposure to one or more Janus Kinase inhibitors (JAKi),[the most recent of which was discontinued > 14 days prior to Cycle 1 Day 1] and are intolerant, resistant, refractory or lost response to the JAKi.
* Segment B:

  * Currently receiving ruxolitinib AND
  * Willingness to reduce ruxolitinib dose (if on a higher dose); and on a stable dose for 14 days or longer prior to Cycle 1 Day 1; AND
  * At least one of the following criteria (a, b, or c):

    1. >= 24 weeks duration of current ruxolitinib course, with evidence of disease that is resistant, refractory, or has lost response to ruxolitinib therapy;
    2. < 24 weeks duration of current ruxolitinib course with documented resistance, refractories, or loss of response, as defined by any of the following:

       * Appearance of new splenomegaly that is palpable to at least 5 cm below the left costal margin (LCM), in participants with no evidence of splenomegaly prior to the initiation of ruxolitinib.
       * >=100% increase in the palpable distance below the LCM, in participants with measurable spleen distance 5 - 10 cm prior to the initiation of ruxolitinib.
       * >=50% increase in the palpable distance below the LCM, in participants with measurable spleen > 10 cm prior to the initiation of ruxolitinib.
       * A spleen volume increase >= 25% (as assessed by MRI or CT) in participants with a spleen volume assessment available prior to the initiation of ruxolitinib.
    3. Prior treatment with ruxolitinib for >= 28 days complicated by any of the following:

       * Development of red blood cell transfusion requirement (at least 2 units/month for 2 months).
       * Grade >= 3 adverse events of neutropenia and/or anemia while on ruxolitinib treatment, with improvement or resolution upon dose reduction.
* Segment C:

  * Prior exposure to one or more JAKi (the most recent of which was discontinued > 14 days prior to Cycle 1 Day 1), and are intolerant, resistant, refractory or lost response to the JAKi.

Exclusion Criteria:

Segment-Specific Prior Therapy Criteria:

* Segment A:

  * Prior exposure to one or more Bromodomain and Extra-Terminal (BET) inhibitors.
* Segment B:

  * Prior exposure to one or more BET inhibitors.
* Segment C:

  * Prior exposure to one or more BET inhibitors and/or any B-Cell Lymphoma 2 (BCL)-2 and/or BCL- XL inhibitor, including navitoclax.
* Segment D:

  * Prior exposure to JAKi and/or any BET inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Up to Approximately 1 year from start of study
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Percentage Of Participants Who Achieve Spleen Volume Reduction Of 35% Or Greater (SVR35) | Up To Week 24
  Reduction in spleen volume is measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
Maximum Observed Plasma Concentration (Cmax) of ABBV-744 | Up To Week 12
  Maximum observed plasma concentration (Cmax) of ABBV-744.
Time To Cmax (Tmax) Of ABBV-744 | Up To Week 12
  The amount of time taken to reach Cmax.
Area Under The Concentration Versus Time Curve (AUC) Of ABBV-744 | Up To Week 12
  AUC of ABBV-744 will be calculated.
Half-Life (t1/2) Of ABBV-744 | Up To Week 12
  Half-life of ABBV-744 will be calculated.
Accumulation Ratio Of ABBV-744 | Up To Week 12
  Pharmacokinetic parameters will include accumulation ratio of ABBV-744.
Apparent Clearance (CL/F) Of ABBV-744 | Up To Week 12
  CL/F of ABBV-744 will be calculated.
Apparent Volume Of Distribution (Vd/F) Of ABBV-744 | Up To Week 12
  Vd/F of ABBV-744 will be calculated.
Percentage Of Participants With >= 50% Reduction In Total Symptom Score (TSS) | Up to Week 24
  TSS is assessed using the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0. MFSAF v4.0 measures the burden of myelofibrosis-related symptoms. The symptoms are assessed on a 11-point numeric rating scale (NRS) anchored from 0 (absent) to 10 (worst imaginable).
Objective Response Rate (ORR) | Week 24
  ORR is defined as the sum of rates of partial remission (PR) or better.
Maximum Observed Plasma Concentration (Cmax) Of Navitoclax | Up To Week 12
  Maximum Observed Plasma Concentration (Cmax) Of Navitoclax.
Time To Cmax (Tmax) Of Navitoclax | Up To Week 12
  The amount of time taken to reach Cmax.
Area Under The Concentration Versus Time Curve (AUC) Of Navitoclax | Up To Week 12
  AUC of Navitoclax will be calculated.
Maximum Observed Plasma Concentration (Cmax) Of Ruxolitinib | Up To Week 12
  Maximum Observed Plasma Concentration (Cmax) Of Ruxolitinib.
Time To Cmax (Tmax) Of Ruxolitinib | Up To Week 12
  The amount of time taken to reach Cmax.
Area Under The Concentration Versus Time Curve (AUC) Of Ruxolitinib | Up To Week 12
  AUC of Ruxolitinib will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (43):
- United States (10):
  - University of California, Davis Comprehensive Cancer Center /ID# 221790, Sacramento, California
  - Duplicate_Dartmouth-Hitchcock Medical Center - 1 Medical Center Drive /ID# 224623, Lebanon, New Hampshire
  - Roswell Park Cancer Institute /ID# 222557, Buffalo, New York
  - The Mount Sinai Hospital /ID# 221549, New York, New York
  - Weill Cornell Medical College /ID# 227069, New York, New York
  - Gabrail Cancer Center Research /ID# 222802, Canton, Ohio
  - University of Oklahoma, Stephenson Cancer Center /ID# 224095, Oklahoma City, Oklahoma
  - Oregon Health and Science University /ID# 221801, Portland, Oregon
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 240004, Dallas, Texas
  - VA Puget Sound Health Care System /ID# 224208, Seattle, Washington
- Argentina (2):
  - Hospital Universitario Austral /ID# 228909, Pilar, Buenos Aires
  - Hospital Italiano de Buenos Aires /ID# 226945, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
- Australia (3):
  - Townsville University Hospital /ID# 225859, Douglas, Queensland
  - Royal Hobart Hospital /ID# 241677, Hobart, Tasmania
  - Royal Perth Hospital /ID# 241678, Perth, Western Australia
- Brazil (6):
  - Hospital das Clinicas da Universidade Federal de Goiás /ID# 226636, Goiânia, Goiás
  - Hospital de Clinicas de Porto Alegre /ID# 226635, Porto Alegre, Rio Grande do Sul
  - Duplicate_Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein /ID# 226640, São Paulo, São Paulo
  - Instituto Nacional de Cancer (INCA) /ID# 226637, Rio de Janeiro
  - Real e Benemérita Associação Portuguesa de Beneficência /ID# 226641, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 226639, São Paulo
- Bulgaria (2):
  - SHAT Hematologic Diseases /ID# 226007, Sofia
  - UMHAT Sveta Marina /ID# 226681, Varna
- Chile (3):
  - Duplicate_Sociedad de Investigaciones Médicas Limitada /ID# 224175, Temuco, Región de la Araucanía
  - Icegclinic /Id# 231086, La Florida, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez /ID# 225037, Providencia, Santiago Metropolitan
- Hungary (2):
  - Clinexpert Kft. Fazis I Vizsgalohely /ID# 242249, Gyöngyös, Heves County
  - Duplicate_Semmelweis Egyetem /ID# 224085, Budapest
- Israel (3):
  - Hadassah Medical Center-Hebrew University /ID# 243852, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 222151, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 223548, Tel Aviv, Tel Aviv
- Duplicate_Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 244397, Milan, Milano, Italy
- Japan (4):
  - Kyushu University Hospital /ID# 228035, Fukuoka, Fukuoka
  - Duplicate_Hokkaido University Hospital /ID# 228038, Sapporo, Hokkaido
  - Osaka Metropolitan University Hospital /ID# 225502, Osaka, Osaka
  - University of Yamanashi Hospital /ID# 225503, Chuo-shi, Yamanashi
- Duplicate_Inje University Busan Paik Hospital /ID# 233707, Busan, Busan Gwang Yeogsi, South Korea
- Spain (2):
  - Hospital Santa Creu i Sant Pau /ID# 238501, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 233279, Madrid
- Sweden (2):
  - Akademiska Sjukhuset /ID# 228515, Uppsala, Uppsala County
  - Orebro Universitetssjukhuset /ID# 228514, Örebro, Örebro County
- Turkey (Türkiye) (2):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi /ID# 234215, Ankara
  - Koc Universitesi Hastanesi Translasyonel Tıp Arastırma Merkezi /ID# 234214, Istanbul

IPD SHARING:
Plan to Share IPD: No